CLINICAL TRIAL: NCT01530061
Title: The Satiating Effect of Eggs in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Egg Nutrition Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PBRC 12001
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Appetite
MeSH Terms: interventions — Eggs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preschool Children age 4-6 years (Experimental): Preschool children participate in eating either an egg breakfast or a bagel breakfast.
  Interventions: Other: Egg Breakfast; Other: Bagel Breakfast
- Teenagers 14-17 years of age (Experimental): Teenagers participate in eating either an egg breakfast or a bagel breakfast.
  Interventions: Other: Egg Breakfast; Other: Bagel Breakfast

INTERVENTIONS:
Other: Egg Breakfast — Egg, Toast and Jelly
  Other Names: Egg
Other: Bagel Breakfast — Bagel, Cream Cheese and Yogurt
  Other Names: Bagel

SUMMARY:
This study will determine which breakfast (egg breakfast or bagel breakfast) has the most beneficial effect on appetite.

DETAILED DESCRIPTION:
Test Day 1 (about 4 hours)

* This is a fasting visit (nothing besides water 12 hours prior to visit)
* Your child will be offered one of two breakfasts (egg breakfast or bagel breakfast)

  . He/she will be asked to eat all the food that is provided.
* He/she will be asked to rate the taste of the meal.
* He/she will be offered a pasta lunch.

Test Day 2 (about 4 hours)

* This will be scheduled 1 week after Test Day 1
* This is a fasting visit (nothing besides water 12 hours prior to visit)
* The procedures for this visit are the same as for Test Day 1. Your child will be offered the breakfast that he/she did not receive at the last visit.

The sequence of the 2 breakfasts will be randomly assigned to each child.

ELIGIBILITY:
Inclusion Criteria:

* • Is a healthy boy or girl between 14 and 17 years of age

  * Is a healthy boy or girl between 4 and 6 years of age

Exclusion Criteria:

* • Is suffering from any diseases such as major heart conditions, type 1 diabetes, cancer, eating disorders, or any serious illness that requires intensive and long-term medical treatment

  * Has allergies/sensitivities/dislikes to eggs, soy, or wheat
  * Uses drugs recreationally
  * Is actively attempting to lose weight

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2012-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Lunch time food intake | 1 day
  Measure calories consumed at lunch time.

SECONDARY OUTCOMES:
Visual Analog Scale Ratings | 1 day
  They will be asked to rate their feelings of hunger and fullness periodically using visual analog scales. The Egg Breakfast is expected to increase satiety scores, decrease hunger and the lunch time food intake, compared to the Bagel Breakfast.
Blood appetite hormone | 1 day
  We expect that Peptide YY (PYY) and Glucagon-like Peptide-1 (GLP1) levels will rise higher and remain elevated after the Egg Breakfast, and the acylated ghrelin levels will rise higher between the Bagle Breakfast and lunch time.

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Dhurandhar, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States